CLINICAL TRIAL: NCT01856868
Title: An Open-label Pilot Study of Purified Tea-derived Epicatechin to Improve Mitochondrial Function, Strength and Skeletal Muscle Exercise Response in Becker Muscular Dystrophy.
Brief Title: Use of (-)-Epicatechin in the Treatment of Becker Muscular Dystrophy (Pilot Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig McDonald, MD (Other)
Collaborators: Cardero Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Craig McDonald, MD, Professor and Chairman, Department of Physical Medicine and Rehabilitation, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 454352
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Becker Muscular Dystrophy
Keywords: BMD; Becker muscular dystrophy; epicatechin; clinical trial; neuromuscular disease
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases | interventions — Catechin; Dietary Supplements

ARMS (1):
- Treatment with Epicatechin (Experimental): Purified nutritional extract (-)-epicatechin 100mg/day orally for 8 weeks.
  Interventions: Drug: (-)-epicatechin

INTERVENTIONS:
Drug: (-)-epicatechin — purified nutritional extract (-)-epicatechin 100mg/day orally for 8 weeks.
  Other Names: dietary supplement

SUMMARY:
(-)-Epicatechin will be evaluated for the treatment of progressive muscle loss and impaired skeletal muscle function in Becker Muscular Dystrophy (BMD) patients.

DETAILED DESCRIPTION:
This is a proof-of-concept phase 1/2a pilot and endpoint development study that is designed to provide initial evidence of biological activity of (-)-epicatechin. Primary endpoints include initial assessment of tissue-specific evidence of efficacy from muscle biopsy samples. Secondary endpoints include measures of strength and physical function, and safety and adverse event data. Pilot endpoints include assessment of mRNA and miRNA peripheral blood profiles and validation of non-invasive near-infrared spectroscopy (NIRS) muscle perfusion studies during exercise and a recumbent cycle exercise test that may be employed as endpoints in future clinical trials.

This single center open-label pilot study will enroll 10 adults with genetically-confirmed Becker muscular dystrophy, who will receive the purified nutritional extract (-)-epicatechin 100mg/day orally for 8 weeks. After screening visits, participants will be enrolled in the study if they meet all inclusion criteria. They will be evaluated at baseline and at screening, day 1, and weeks 1, 2, 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 years to 60 years
* Average to low daily physical activity
* Ability to ambulate for 75 meters without assistive devices
* Diagnosis of BMD confirmed by at least one the following:

  * Dystrophin immunofluorescence and/or immunoblot showing partial dystrophin deficiency, and clinical picture consistent with typical BMD, or
  * Gene deletions test positive (missing one or more exons) of the dystrophin gene, where reading frame can be predicted as 'in-frame', and clinical picture consistent with typical BMD, or
  * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, or other mutation resulting in a stop codon mutation) that can be definitely associated with BMD, with a typical clinical picture of BMD, or
  * Positive family history of BMD confirmed by one of the criteria listed above in a sibling or maternal uncle, and clinical picture typical of BMD.
* Nutritional, herbal and antioxidant supplements taken with the intent of maintaining or improving skeletal muscle strength or functional mobility have been discontinued at least 2 weeks prior to screening (daily multivitamin use is acceptable).
* Hematology profile within normal range
* Baseline laboratory safety chemistry profile within normal range
* No plan to change exercise regimen during study participation

Exclusion Criteria:

* Currently enrolled in another treatment clinical trial.
* History of significant concomitant illness or significant impairment of renal or hepatic function.
* Use of regular daily aspirin or other medication with antiplatelet effects within 3 weeks of first dose of study medication.
* Regular participation in vigorous exercise.
* Symptomatic heart failure with cardiac ejection fraction <25%

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig M McDonald, MD, Principal Investigator — University of California, Davis; Erik K Henricson, MPH, Study Director — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- See also: UC Davis Neuromuscular Research Center — http://www.ucdmc.ucdavis.edu/pmr/research/Index.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Epicatechin
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 179.2 (4.3)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 83.2 (18.3)
Forced Vital Capacity (%) [Mean (Standard Deviation); unit: %] | 93.4 (12.5)
6-Minute Walk Distance (m) [Mean (Standard Deviation); unit: meters] | 372 (87.2)
Time to Stand (s) [Mean (Standard Deviation); unit: seconds] | 5.5 (2.3)
Time to Climb 4 Stairs (s) [Mean (Standard Deviation); unit: seconds] | 7.4 (7.4)
Time to Run 10m (s) [Mean (Standard Deviation); unit: seconds] | 7.9 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Muscle Tissue PGC1alpha (AU) at 8 Weeks
Description: Western blot measurement of the transcriptional coactivator gene PGC1alpha involved in mitochondrial biogenesis will be assessed using relative band intensities of the pre-treatment (Baseline) and post-treatment (8 Weeks) specimens with digitally quantified using ImageJ software.
Time Frame: Baseline and 8 Weeks
Population: One participant sustained a fall at home that resulted in a minor injury just prior to the 8 week evaluation and declined undergoing the 8 week biopsy. Thus, only 6 participants were analyzed.
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.55 (0.3)
  8 Weeks | 0.86 (0.17)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0434, t-test, 2 sided

2. Primary Outcome: Mean Change From Baseline in Muscle Tissue AMPK at 8 Weeks
Description: Western blot measurement of AMPK will be assessed using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.76 (0.48)
  Week 8 | 1.06 (0.52)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0185, t-test, 2 sided

3. Primary Outcome: Mean Change From Baseline in Muscle Tissue LKB1 at 8 Weeks
Description: Western blot measurement of LKB1 will be assessed using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software) .
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.67 (0.17)
  Week 8 | 0.88 (0.24)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0434, t-test, 2 sided

4. Primary Outcome: Mean Change From Baseline in Cristae-associated Mitofillin Levels at 8 Weeks
Description: Western blot measurement of Mitofillin will be assessed using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 1.05 (0.36)
  Week 8 | 1.33 (0.3)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0078, t-test, 2 sided

5. Primary Outcome: Mean Change From Baseline in Muscle Tissue Follistatin at 8 Weeks
Description: Regulators of muscle growth and regeneration including follistatin will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.83 (0.37)
  Week 8 | 1.11 (0.36)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0025, t-test, 2 sided

6. Primary Outcome: Mean Change From Baseline in Muscle Tissue Myostatin at 8 Weeks
Description: Regulators of muscle growth and regeneration including myostatin will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.79 (0.3)
  Week 8 | 0.51 (0.25)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0082, t-test, 2 sided

7. Primary Outcome: Mean Change From Baseline in Muscle Tissue Myogenin at 8 Weeks
Description: Modulators of skeletal muscle regeneration by Western will include myogenin will be assessed using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.89 (0.18)
  Week 8 | 1.20 (0.19)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.031, t-test, 2 sided

8. Primary Outcome: Mean Change From Baseline in Muscle Tissue Myf5 at 8 Weeks
Description: Modulators of skeletal muscle regeneration My5 will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 1.07 (0.08)
  Week 8 | 1.232 (0.13)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0238, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Mean Change From Baseline in Muscle Tissue MyoD at 8 Weeks
Description: Modulators of skeletal muscle regeneration MyoD will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.87 (0.34)
  Week 8 | 1.21 (0.34)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0321, t-test, 2 sided

10. Primary Outcome: Mean Change From Baseline in Muscle Tissue MEF2a at 8 Weeks
Description: Modulators of skeletal muscle regeneration MEF2a will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.63 (0.15)
  Week 8 | 0.78 (0.12)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0182, t-test, 2 sided

11. Primary Outcome: Mean Change From Baseline in Muscle Tissue Dysferlin at 8 Weeks
Description: Structure associated indicators including dysferlin will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.65 (0.26)
  Week 8 | 0.91 (0.25)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0371, t-test, 2 sided

12. Primary Outcome: Mean Change From Baseline in Muscle Tissue Utrophin at 8 Weeks
Description: Structure associated indicators including utrophin will be assessed by Western using relative band intensities of the pre-treatment and post-treatment specimens with digitally quantified using ImageJ software).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
AU
  Baseline | 0.63 (0.27)
  Week 8 | 0.8 (0.19)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a paired t-test analysis; p = 0.0257, t-test, 2 sided

13. Secondary Outcome: -(-)Epicatechin Pharmacokinetics
Description: Pharmacokinetics sequentially after dosing will be measured.
Time Frame: 8 Weeks
Population: Sponsor did not perform PK analysis (samples were discarded) based on availability of other published data and switched to alternative enantiomer of epicatechin in subsequent studies.
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 0

14. Secondary Outcome: Participants With Abnormal Treatment-Related Laboratory Assessments
Description: Standard safety monitoring of plasma hematologic, hepatologic, renal and metabolic parameters will be assessed. Abnormal will be defined as values outside of typical range for patients with Becker Muscular Dystrophy.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 7
Participants | 0

15. Secondary Outcome: Change From Baseline in Knee Extension at 8 Weeks
Description: Knee extension will be assessed using an isokinetic dynamometer.
Time Frame: Baseline and 8 Weeks
Population: One participant did not participate in the strength testing due to the advanced level of the disease.
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
pounds
  Baseline | 48.1 (42.6)
  Change from Baseline at 8 Weeks | -1.82 (2.51)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a mixed model regression analysis, including fixed effects for height and weight using patient identity as source of random variation. As a pilot study, these measures were not subject to a formal power analysis but will be used in future sample size calculations; p = 0.47, Mixed Models Analysis; Mean Difference (Net) = -1.82, Standard Error of Mean 2.51

16. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance at 8 Weeks
Description: Muscle function will be assessed by measuring the 6-minute walk distance
Time Frame: Baseline and 8 Weeks
Population: One participant did not complete 8 Week exercise testing due to unrelated injury.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
meters | 11.2 (16.6)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — Difference in baseline and 8 week scores was evaluated using a mixed model regression analysis, including fixed effects for height, weight and knee extension strength using patient identity as source of random variation. As a pilot study, these measures were not subject to a formal power analysis but will be used in future sample size calculations; p = 0.50, Mixed Models Analysis; Mean Difference (Net) = 11.2, Standard Error of Mean 16.6

17. Secondary Outcome: Change From Baseline in Stand From Supine at 8 Weeks
Description: Muscle burst function will be assessed by time function tests.
Time Frame: Baseline and 8 Weeks
Population: 1 participant was unable to perform the assessment due to his advanced disease.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
seconds
  Baseline | 9.621667 (10.19124)
  Week 8 | 12.145 (10.12084)

18. Secondary Outcome: Change From Baseline in Elbow Flexion at 8 Weeks
Description: Elbow flexion will be assessed using an isokinetic dynamometer.
Time Frame: Baseline and 8 Weeks
Population: One participant did not participate in the strength testing due to the advanced level of the disease.
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Treatment With Epicatechin
Number analyzed (Participants) | 6
pounds
  Baseline | 27.7 (11.1)
  Change from Baseline at 8 Weeks | 5.33 (3.79)
Statistical Analysis 1: Comparison: Treatment With Epicatechin; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.159, Mixed Models Analysis; Mean Difference (Net) = 5.33, Standard Error of Mean 3.79

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: There were 12 adverse events in six participants reported and tracked during the 8-week treatment phase of the study. Seven of the 12 events were related or possibly related to the study biopsy procedure. All adverse events were followed until resolution.
Arm/Group | Treatment With Epicatechin
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Epicatechin (N=6)
Bruising at the biopsy site (Skin and subcutaneous tissue disorders) | 6 (6)
Non-biopsy-related flulike symptoms (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
suspected varicella (shingles) (Immune system disorders) | 1 (1)
Muscle soreness (General disorders) | 1 (1)
Intermittent headache (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study include the small number of subjects, the open-label design, and the use of within-subjects controls with BMD rather than a placebo-treated group in a randomized, double-blind, placebo-controlled trial design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-03-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT01856868/Prot_SAP_000.pdf
  • Informed Consent Form (2014-03-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT01856868/ICF_001.pdf